CLINICAL TRIAL: NCT02551211
Title: Association Between Circulating Immune Cells and the Tumor Immune Contexture in Resectable Non-small Cell Lung Cancer
Acronym: LYMPHOLUNG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: 2015/080/HP
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Resectable Non-small Lung Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with resectable non-small cell lung cancer (Experimental)
  Interventions: Procedure: blood drawn; Procedure: surgical resection of cancer

INTERVENTIONS:
Procedure: blood drawn — blood drawn
Procedure: surgical resection of cancer

SUMMARY:
With the recent approval of Nivolumab for second-line treatment of stage IIIb/IV non-small cell lung cancer (NSCLC), immune checkpoint inhibitors are entering the standard of care for lung cancer. Other immune checkpoint inhibitors are under evaluation, both in resectable and non-resectable NSCLC. In order to refine our use of these molecules, comprehensive data on the immune contexture of NSCLC are needed. Moreover,a blood marker of this contexture would allow physicians to monitor the immune status of their patient's tumor and though to evaluate the rightful place of immunotherapy in the multimodal treatment of NSCLC. No such blood marker has been validated so far. The LYMPHOLUNG study investigate the concordance between blood and intratumoral counts of immune cells in resectable stage I to IIIA NSCLC. By the use of 30-marker cytometry, a precise immune profile of NSCLC will be depicted. The prognostic value of the circulating and intra-tumoral T regulator over total lymphocytes ratio for 2-year recurrence-free survival will also be addressed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age
* Histologically- or cytologically- confirmed non-small cell lung cancer diagnostic
* Stage I, II or IIIA NSCLC (according to version 7 of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology). Staging must have included an abdominal and thoracic CTscan, a CTscan or MRI of the brain and a 18FDG PETscan
* Subjects for whom a surgical resection is indicated
* Signed written informed consent

Exclusion Criteria:

* - previous, ongoing or planned neo-adjuvant treatment (chemotherapy, targeted therapy, immunotherapy or radiotherapy)
* contraindications to general anesthesia
* contraindication to the planned surgical resection
* history of immunosuppressive disorder
* known history of testing positive for human immunodeficiency virus
* subjects with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 30 days of randomization.
* clinical suspicion of active infection (either acute or chronic)
* severe (hemoglobin < 8.0 g/dL) or symptomatic anemia
* women of childbearing potential must have a negative urine pregnancy test
* women must not be breastfeeding
* prisoners or subjects who are involuntarily incarcerated
* subjects under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Level of expression of the T regulator over total lymphocytes count ratio in the blood | Day 1
Level of expression of the T regulator over total lymphocytes count ratio into the tumor | Day 1

SECONDARY OUTCOMES:
Number of cell population counts as blood markers for the corresponding population in the tumor | Day 1
Number of patient alive 2 years after resection | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bérengère OBSTOY, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France